CLINICAL TRIAL: NCT06457724
Title: Randomized Controlled Trial on the Effect of Levilactobacillus Brevis (CNCM I-5566) Probiotic Supplement on Clinical and Salivary Oral Indicators
Brief Title: Levilactobacillus Brevis Oral Health
Acronym: LBOH-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Davide Pietropaoli, Associate Professor, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 48/2022
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Oral Health; Oral Disease
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L. brevis (Experimental)
  Interventions: Dietary Supplement: Levilactobacillus brevis CNCM I-5566
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Levilactobacillus brevis CNCM I-5566 — Participants will take four Mucomixx tablets (containing Levilactobacillus brevis CNCM I-5566) daily for 28 days. The tablets should be taken after each of the following meals: breakfast, lunch, afternoon break, and dinner.
  Other Names: Mucomixx
  Arms: L. brevis
Dietary Supplement: Placebo — Participants will take four placebo tablets daily for 28 days. The tablets should be taken after each of the following meals: breakfast, lunch, afternoon break, and dinner.
  Arms: Placebo

SUMMARY:
This RCT investigates the impact of an oral supplement containing the probiotic Levilactobacillus brevis CNCM I-5566 on various salivary indicators of oral health. Participants will be randomly assigned to either the probiotic supplement group or a placebo group. The primary objective is to assess changes in salivary biomarkers, including salivary pH and buffer capacity; microbial composition using microbiome next-generation sequencing (NGS); and clinical oral inflammatory markers, such as full mouth bleeding score and full mouth plaque score, over a 4-week period. By comparing these indicators between the two groups, the study aims to determine the efficacy of Levilactobacillus brevis CNCM I-5566 in promoting oral health and potentially preventing oral diseases.

DETAILED DESCRIPTION:
This RCT is designed to investigate the impact of an oral supplement containing the probiotic Levilactobacillus brevis CNCM I-5566 on various salivary indicators of oral health. The study aims to provide robust evidence on the efficacy of this probiotic in promoting oral health and potentially preventing oral diseases.

Study Design:

Participants will be randomly assigned to one of two groups: the experimental group, which will receive the Levilactobacillus brevis CNCM I-5566 probiotic supplement, and the control group, which will receive a placebo. This random assignment ensures that the groups are comparable at the start of the trial, allowing for unbiased comparison of outcomes.

Duration:

The study will be conducted over a 4-week treatment period, during which participants will adhere to their assigned supplement regimen.

Primary Objectives:

The primary objective of this RCT is to assess the impact of Levilactobacillus brevis CNCM I-5566 on several key indicators of oral health, measured through salivary biomarkers, microbial composition, and clinical oral inflammatory markers.

Salivary Biomarkers:

Salivary pH: The acidity or alkalinity of saliva, which can influence oral health by affecting the growth of bacteria and the integrity of tooth enamel.

Buffer Capacity: The ability of saliva to neutralize acids, which is crucial for maintaining a healthy oral environment and preventing dental caries.

Salivation rate: The amount of salivary production (mL) overtime (in 5 minutes). This parameter is needed for individual caries risk assessment.

Microbial Composition:

The composition of the oral microbiome will be analyzed using next-generation sequencing (NGS). This advanced technique allows for a comprehensive assessment of the microbial populations present in the saliva and dental plaque, providing insights into how the probiotic supplement may alter the microbiome to support oral health.

Clinical Oral Inflammatory Markers:

Full Mouth Bleeding Score: A measure of gum inflammation and bleeding, which are indicators of gingivitis or periodontal disease.

Full Mouth Plaque Score: A measure of the accumulation of dental plaque, which is a biofilm of bacteria that can lead to tooth decay and gum disease if not properly managed.

Outcome Comparison:

By comparing the changes in these indicators between the probiotic supplement group and the placebo group, the study aims to determine the efficacy of Levilactobacillus brevis CNCM I-5566. Significant improvements in the probiotic group compared to the placebo group would suggest that Levilactobacillus brevis CNCM I-5566 is effective in promoting oral health and preventing oral diseases.

Significance:

This study has the potential to contribute valuable information to the field of oral health, particularly in understanding how probiotics can be used as a preventive measure against oral diseases. If successful, the findings could lead to new recommendations for probiotic use in dental care routines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes.
* Dental caries experience (DMFT) less than 4.

Exclusion Criteria:

* Active or historical periodontitis.
* Diabetes mellitus diagnosis.
* Active or historical cancer diagnosis.
* Antibiotic therapy within the past 3 months.
* Currently undergoing active therapy with drugs.
* Presence of disabilities affecting the ability to maintain oral hygiene at home.
* Recent professional oral hygiene treatment within the last 3 months.
* Pregnancy.
* Presence of eating disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Salivary pH | Baseline, 4 and 6 weeks
  Assay used to define dental caries risk
Full mouth bleeding score | Baseline, 4 and 6 weeks
  Index used to quantify gingival inflammation (Percentage as Full mouth Bleeding score)
Full mouth plauqe score | Baseline, 4 and 6 weeks
  Index used to quantify individual capacity to home oral health (Percentage as Full mouth Plaque score)

CONTACTS AND LOCATIONS:
Locations (1):
- University of L'Aquila, L’Aquila, IT, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Altamura S, Lombardi F, Augello FR, Barone A, Giannoni M, Cinque B, Pietropaoli D. Levilactobacillus brevis CD2 as a multifaceted probiotic to preserve oral health: results of a double-blind, randomized, placebo-controlled trial in healthy adults. J Transl Med. 2025 Jan 28;23(1):128. doi: 10.1186/s12967-024-06000-1. PMID 39875908